CLINICAL TRIAL: NCT04424628
Title: Three vs Six Gy in Gonarthrosis and Coxarthrosis. Non Inferiority Study
Brief Title: Radiotherapy 3 vs 6 Gy in Gonarthrosis and Coxarthrosis
Acronym: RAGOCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion GenesisCare (Network)
Collaborators: Elekta Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GEN-RAD-2019-01
Record Dates: First submitted 2020-06-01; First posted 2020-06-11 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Gonarthrosis; Coxarthrosis
Keywords: Low Dose Radiotherapy; Anti-inflammatory effects; Pain release; Quality of Life
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Arm 1: 3 Gy (repeated at 8 weeks if necessary. New ramdomization to 3 Gy or 6 Gy) Arm 2: 6 Gy (repeated at 8 weeks if necessry)
Who Masked: Participant
Masking Description: Patients label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy 3 Gy (Active Comparator): Patiens will receive low dose gonarthrosis or coxarthrosis radiotherapy (0.5 Gy in 6 fractions alternating days).
  Evaluation of pain releave and quality of live in 8-12 weeks If no effect the patient will be randomized to 3 or 6 Gy again
  Interventions: Radiation: Low dose radiotherapy A
- Radiotherapy 6 Gy (Active Comparator): Patiens will receive low dose gonarthrosis or coxarthrosis radiotherapy (1 Gy in 6 fractions alternating days).
  Evaluation of pain releave and quality of live in 8-12 weeks If no effect the patient will be treated with 6 Gy again
  Interventions: Radiation: Low dose radiotherapy B

INTERVENTIONS:
Radiation: Low dose radiotherapy A — Low dose radiotherapy was 0.5 Gy in 6 fractions. Evaluation of pain and Quality of Life in 8-12 weeks. If no pain releave the patient is randomized to 3 or 6 Gy again
  Arms: Radiotherapy 3 Gy
Radiation: Low dose radiotherapy B — Low dose radiotherapy was 0.5 Gy in 6 fractions. Evaluation of pain and Quality of Life in 8-12 weeks. If no pain releave the patient is treated with 6 Gy again
  Arms: Radiotherapy 6 Gy

SUMMARY:
This is a non-inferiority study in which the investigators compare two low-dose radiotherapy schemes, which are recommended from DEGRO Clinical Practice Guidelines (3 Gy vs 6 Gy) for the treatment of osteoarthritis and other osteodegenerative disorders.

A first randomization will be carried out among the patients included in the study:

* Patients in arm A will be treated at 3 Gy (0.5 Gy/fraction, 3 fractions/week), and patients in arm B will be treated at 6 Gy (1 Gy/fraction, 3 fractions/week).
* Patients should not know the arm to which they have been randomized.
* Once the treatment is finished, patients will be assessed at 8 weeks. If pain does not improve, a re-irradiation will be performed. If the patients were treated with 3 Gy a new randomization will be performed (3 vs 6 Gy again). If the patiens were treated with 6 Gy they will be re-irradiated with 6 Gy again.

The investigators will analyze the results obtained depending on the dose received and depending on the location of the treatment.

DETAILED DESCRIPTION:
Painfull skeletal disorders are susceptible to be treated with low-dose radiotherapy. DEGRO guidelines recommend a dose between 3 and 6 Gy at 0'5 Gy/fraction or 1 Gy/fraction respectively. The investigators want to verify that both treatments (3 and 6 Gy) are similar to improve the pain and function in patiens with gonarthrosis and coxarthrosis, and there are no differences between both treatments, therefore, 3 Gy is not less than 6 Gy.

In this context, a prospective multicenter study is proposed. The study will include 338 patients to assess the efficacy of low dose irradiation (3 vs 6 Gy) in gonarthrosis and coxarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years
* Gonarthrosis or/and Coxarthrosis diagnose
* At least 1 year of evolution
* Non response to drug or surgery treatments
* Risk of colateral side effects due to the comorbidity of the patient with conventional treatments.

Exclusion Criteria:

* Previous high dose radiotherapy in the same location
* Conective tissue disease (LUPUS, reumathoid artritis, esclerodermia, Sd. Raynaud, Sd. Sjögren, polymiositis)
* Inherited Hipersesitivity Sindromes (ataxia-telangiectasia, Fanconi's anaemya, Sd. Nijmegen, Sd. Gorlyn, Sd. Cockayne, Sd. Down, Sd. Gardner, Sd. Usher)
* No follow up possibility
* Other study inclusion

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain control at 8-12 weeks and every 6 months | At 8-12 weeks, 6 months, 12 months, 18 months and 24 months
  To evaluate the non inferiority efficacy of low dose radiotherapy 3 or 6 Gy to change in pain with VAS (Visual Analogue Scale). The patient scores his painfrom 0 (no hurt) to 10 (hurts worst). It is better a low score.
Quality of Life at 8-12 weeks and every 6 months | At 8-12 weeks, 6 months, 12 months, 18 months and 24 months
  To evaluate the non inferiority efficacy of low dose radiotherapy 3 or 6 Gy to change in pain with WOMAC scale (Western Ontario MacMaster Questionnaire). This questionnaire has 24 questions about pain, joint stiffness and joint function. It is better a low score.

SECONDARY OUTCOMES:
Skin toxicity at 8-12 weeks. | At 8-12 weeks.
  Skin toxicity will be assessed and rated acording to the RTOG scale (0= no change over baseline; 1: Follicular, faint or dull erythema epilation, dry desquamation, decreased sweating; 2: Tender or bright erythema, patchy moist desquamation, moderate oedema; 3: Confluent, moist desquamation other tan skin folds, pitting oedema; 4: Ulceration haemorrhege, necrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rivas Sanchez, MD, Principal Investigator — Fundacion GenesisCare
Locations (1):
- GenesisCare Malaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No
The overall results of any research conducted Will be available on study data publication
  Supportin information:
  Study protocol Informed Consent Form (ICF)

REFERENCES:
- [Background] Micke O, Seegenschmiedt MH; German Working Group on Radiotherapy in Germany. Consensus guidelines for radiation therapy of benign diseases: a multicenter approach in Germany. Int J Radiat Oncol Biol Phys. 2002 Feb 1;52(2):496-513. doi: 10.1016/s0360-3016(01)01814-4. PMID 11872298
- [Background] Montero Luis A, Hernanz de Lucas R, Hervas Moron A, Fernandez Lizarbe E, Sancho Garcia S, Vallejo Ocana C, Polo Rubio A, Ramos Aguerri A. Radiation therapy for the treatment of benign vascular, skeletal and soft tissue diseases. Clin Transl Oncol. 2008 Jun;10(6):334-46. doi: 10.1007/s12094-008-0209-6. PMID 18558580
- [Background] Reichl B, Block A, Schafer U, Bert C, Muller R, Jung H, Rodel F; German Cooperative Group on Radiotherapy for Benign Diseases (GCG-BD). DEGRO practical guidelines for radiotherapy of non-malignant disorders: Part I: physical principles, radiobiological mechanisms, and radiogenic risk. Strahlenther Onkol. 2015 Sep;191(9):701-9. doi: 10.1007/s00066-015-0865-8. Epub 2015 Jun 28. PMID 26117368
- [Background] Smith-Bindman R, Lipson J, Marcus R, Kim KP, Mahesh M, Gould R, Berrington de Gonzalez A, Miglioretti DL. Radiation dose associated with common computed tomography examinations and the associated lifetime attributable risk of cancer. Arch Intern Med. 2009 Dec 14;169(22):2078-86. doi: 10.1001/archinternmed.2009.427. PMID 20008690
- [Background] Jansen JT, Broerse JJ, Zoetelief J, Klein C, Seegenschmiedt HM. Estimation of the carcinogenic risk of radiotherapy of benign diseases from shoulder to heel. Radiother Oncol. 2005 Sep;76(3):270-7. doi: 10.1016/j.radonc.2005.06.034. PMID 16157402
- [Background] Minten MJM, Leseman-Hoogenboom MM, Kloppenburg M, Kortekaas MC, Leer JW, Poortmans PMP, van den Hoogen FHJ, den Broeder AA, van den Ende CHM. Lack of beneficial effects of low-dose radiation therapy on hand osteoarthritis symptoms and inflammation: a randomised, blinded, sham-controlled trial. Osteoarthritis Cartilage. 2018 Oct;26(10):1283-1290. doi: 10.1016/j.joca.2018.06.010. Epub 2018 Jul 7. PMID 30231990
- [Background] Arenas M, Sabater S, Hernandez V, Rovirosa A, Lara PC, Biete A, Panes J. Anti-inflammatory effects of low-dose radiotherapy. Indications, dose, and radiobiological mechanisms involved. Strahlenther Onkol. 2012 Nov;188(11):975-81. doi: 10.1007/s00066-012-0170-8. Epub 2012 Aug 22. PMID 22907572
- [Background] Kern PM, Keilholz L, Forster C, Hallmann R, Herrmann M, Seegenschmiedt MH. Low-dose radiotherapy selectively reduces adhesion of peripheral blood mononuclear cells to endothelium in vitro. Radiother Oncol. 2000 Mar;54(3):273-82. doi: 10.1016/s0167-8140(00)00141-9. PMID 10738086
- [Background] Hildebrandt G, Seed MP, Freemantle CN, Alam CA, Colville-Nash PR, Trott KR. Mechanisms of the anti-inflammatory activity of low-dose radiation therapy. Int J Radiat Biol. 1998 Sep;74(3):367-78. doi: 10.1080/095530098141500. PMID 9737539
- [Background] Leer JW, van Houtte P, Davelaar J. Indications and treatment schedules for irradiation of benign diseases: a survey. Radiother Oncol. 1998 Sep;48(3):249-57. doi: 10.1016/s0167-8140(98)00051-6. PMID 9925244
- [Result] Ott OJ, Niewald M, Weitmann HD, Jacob I, Adamietz IA, Schaefer U, Keilholz L, Heyd R, Muecke R; German Cooperative Group on Radiotherapy for Benign Diseases (GCG-BD). DEGRO guidelines for the radiotherapy of non-malignant disorders. Part II: Painful degenerative skeletal disorders. Strahlenther Onkol. 2015 Jan;191(1):1-6. doi: 10.1007/s00066-014-0757-3. Epub 2014 Sep 20. PMID 25238992
- [Result] Seegenschmiedt MH, Katalinic A, Makoski H, Haase W, Gademann G, Hassenstein E. Radiation therapy for benign diseases: patterns of care study in Germany. Int J Radiat Oncol Biol Phys. 2000 Apr 1;47(1):195-202. doi: 10.1016/s0360-3016(99)00537-4. PMID 10758324
- [Result] Leer JW, van Houtte P, Seegenschmiedt H. Radiotherapy of non-malignant disorders: where do we stand? Radiother Oncol. 2007 May;83(2):175-7. doi: 10.1016/j.radonc.2007.04.008. Epub 2007 May 8. PMID 17490769
- [Result] Seegenschmiedt MH. New future for radiation therapy of non-malignant diseases? Radiother Oncol. 2005 Jan;74(1):1-2. doi: 10.1016/j.radonc.2005.01.001. No abstract available. PMID 15683660
- [Result] Micke O, Ugrak E, Bartmann S, Adamietz IA, Schaefer U, Bueker R, Kisters K, Heinrich Seegenschmiedt M, Fakhrian K, Muecke R. Radiotherapy for calcaneodynia, achillodynia, painful gonarthrosis, bursitis trochanterica, and painful shoulder syndrome - Early and late results of a prospective clinical quality assessment. Radiat Oncol. 2018 Apr 19;13(1):71. doi: 10.1186/s13014-018-1025-y. PMID 29673383
- [Result] Kriz J, Seegenschmiedt HM, Bartels A, Micke O, Muecke R, Schaefer U, Haverkamp U, Eich HT. Updated strategies in the treatment of benign diseases-a patterns of care study of the german cooperative group on benign diseases. Adv Radiat Oncol. 2018 Feb 26;3(3):240-244. doi: 10.1016/j.adro.2018.02.008. eCollection 2018 Jul-Sep. PMID 30197936
- [Result] Minten MJ, Mahler E, den Broeder AA, Leer JW, van den Ende CH. The efficacy and safety of low-dose radiotherapy on pain and functioning in patients with osteoarthritis: a systematic review. Rheumatol Int. 2016 Jan;36(1):133-42. doi: 10.1007/s00296-015-3337-7. Epub 2015 Aug 8. PMID 26747050
- [Result] Micke O, Seegenschmiedt MH, Adamietz IA, Kundt G, Fakhrian K, Schaefer U, Muecke R; German Cooperative Group on Radiotherapy for Nonmalignant Diseases (GCG-BD). Low-Dose Radiation Therapy for Benign Painful Skeletal Disorders: The Typical Treatment for the Elderly Patient? Int J Radiat Oncol Biol Phys. 2017 Jul 15;98(4):958-963. doi: 10.1016/j.ijrobp.2016.12.012. Epub 2016 Dec 18. PMID 28258900
- [Result] Koc BB, Schotanus MGM, Borghans R, Jong B, Maassen ME, Buijsen J, Jansen EJP. Short-term pain reduction after low-dose radiotherapy in patients with severe osteoarthritis of the hip or knee joint: a cohort study and literature review. Eur J Orthop Surg Traumatol. 2019 May;29(4):843-847. doi: 10.1007/s00590-019-02377-8. Epub 2019 Jan 16. PMID 30649618
- [Result] Mucke R, Seegenschmiedt MH, Heyd R, Schafer U, Prott FJ, Glatzel M, Micke O; German Cooperative Group on Radiotherapy for Benign Diseases (GCG-BD). [Radiotherapy in painful gonarthrosis. Results of a national patterns-of-care study]. Strahlenther Onkol. 2010 Jan;186(1):7-17. doi: 10.1007/s00066-009-1995-7. Epub 2009 Dec 28. German. PMID 20082182
- [Result] Seegenschmiedt MH, Micke O. [Radiotherapy of non-malignant diseases. Past, present and future]. Strahlenther Onkol. 2012 Nov;188 Suppl 3:272-90. doi: 10.1007/s00066-012-0195-z. No abstract available. German. PMID 23053149
- [Result] Reinartz G, Eich HT, Pohl F; German Cooperative Group on Radiotherapy for Benign Diseases (GCG-BD). DEGRO practical guidelines for the radiotherapy of non-malignant disorders - Part IV: Symptomatic functional disorders. Strahlenther Onkol. 2015 Apr;191(4):295-302. doi: 10.1007/s00066-014-0789-8. Epub 2014 Dec 9. PMID 25487694
- [Result] Keller S, Muller K, Kortmann RD, Wolf U, Hildebrandt G, Liebmann A, Micke O, Flemming G, Baaske D. Efficacy of low-dose radiotherapy in painful gonarthritis: experiences from a retrospective East German bicenter study. Radiat Oncol. 2013 Jan 31;8:29. doi: 10.1186/1748-717X-8-29. PMID 23369282
- [Result] Hautmann MG, Jung EM, Beyer LP, Suss C, Steger F, Weber M, Pohl F, Kolbl O, Putz FJ. Is low dose radiotherapy an effective treatment for Baker's cyst? Strahlenther Onkol. 2019 Jan;195(1):69-76. doi: 10.1007/s00066-018-1389-9. Epub 2018 Oct 30. PMID 30377698